CLINICAL TRIAL: NCT01595997
Title: A Multi-center, Double-blinded, Randomized, Placebo-controlled, Intra-individual Comparison, Phase Ib Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Intra-dermal Injections of DLX105 Into Lesional Skin in Patients With Mild-to-moderate Psoriasis Vulgaris
Brief Title: Intra-dermal Injections of DLX105 Into Lesional Skin in Patients With Mild-to-moderate Psoriasis Vulgaris
Acronym: 2011-00500-15
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Delenex Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLX105-003-001-001
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Mild-to-moderate Psoriasis Vulgaris
Keywords: safety tolerability and immunogenicity of two different doses of DLX105 applied intra-dermally into psoriatic lesion of mild-to-moderate psoriatic patients

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: DLX105
- DLX105 (Experimental)
  Interventions: Drug: DLX105

INTERVENTIONS:
Drug: DLX105 — intradermal injections (volume: 0.1 mL) of 0.02 mg (low dose cohort), 1 mg (high dose cohort) DLX105, days: Day 1, Day 4, Day 7 and Day 10

SUMMARY:
The overall purpose of this study is to support the development of a DLX105 topical formulation for the indication mild to moderate psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent
* Male or female Caucasian patients with stable chronic mild-to-moderate plaque-type psoriasis (PASI ≤15) aged 18-75 years who must have at least two pronounced but not active lesions of >9 cm2 each, stable for at least 3 months, local PASI score ≥8. Distance between lesions must be at least 30 cm.
* Affected body surface area (BSA) ≤10%
* Negative pregnancy test for females of child bearing potential (pre-menopausal, <2 years post-menopausal, not surgically sterile)

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis, palmar, plantar or nail disease) at screening
* Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium) prior to randomization
* Ongoing use of psoriasis treatments (duration of washout, i.e. discontinuation prior to randomization):
* Alefacept (6 months)
* Biological agents other than alefacept, e.g. adalimumab, efalizumab, etanercept, infliximab, ustekinumab (12 weeks)
* Systemic therapy for psoriasis and psoriatic arthritis (other than above) e.g. methotrexate, cyclosporin, fumaric acid (derivatives), systemic steroids (4 weeks)
* Photochemotherapy e.g., ultraviolet A with psoralen (PUVA) (4 weeks)
* Phototherapy e.g., ultraviolet A (UVA) or ultraviolet B (UVB) (2 weeks)
* Topical treatments, except in face, scalp and genital area during screening (2 weeks)
* Other investigational psoriasis drugs (4 weeks or 5 half-lives, whichever is longer)
* Ongoing use of other (non-psoriasis) treatments (duration of washout, i.e. discontinuation prior to randomization):
* Investigational drugs, not psoriasis drugs (4 weeks or 5 half-lives, whichever is longer)
* Known immunosuppression
* History or evidence of active tuberculosis. All patients will be tested for tuberculosis status using a blood test (QuantiFERON TB-Gold) unless this test has been performed within 4 months prior to randomization and was negative. Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment has been initiated according to local regulations.
* Active systemic infections (other than common cold) during the two weeks before randomization
* Positive test for hepatitis B or C at screening
* Positive test for HIV at screening
* History or symptoms of malignancy of any organ system (other than history of basal cell carcinoma and / or up to three squamous cell carcinomas of the skin, if successful treatment has been performed, with no signs of recurrence; actinic keratoses, if present at screening, should be treated according to standard therapy before randomization), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of severe hypersensitivity to any human or humanized biological agents
* Any severe, progressive or uncontrolled medical condition at baseline that in the judgment of the investigator prevents the patient from participating in the study
* Any clinically significant abnormal laboratory tests at baseline
* Active liver disease with alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) > 3 x upper limit of normal
* History of moderate or severe congestive heart failure (New York Heart Association [NYHA] class III or IV).
* Inability or unwillingness to undergo repeated venipunctures (e.g., due to poor tolerability or lack of access to veins)
* History or evidence of drug or alcohol abuse within the 6 months prior first study drug administration
* Patients who had live vaccination within 6 weeks prior first study drug administration, or will require live vaccination during the course of the trial
* History of hypersensitivity to any of the excipients of the study drug or to excipients of similar chemical classes
* History of hypersensitivity to any active ingredient of similar chemical entity (polypeptides)
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (HCG) laboratory test (> 5 mIU/mL)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. UNLESS they are
* Women whose partners have been sterilized by vasectomy or other means
* Using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, condoms (by the partner), and some intrauterine devices (IUDs)). Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered acceptable forms of birth control within this study.
* Reliable contraception should be maintained throughout the study and for 12 weeks after the last study drug administration
* Participation in any other clinical trial within 4 weeks prior to or during this trial
* Exposure to DLX105 / ESBA105 in previous studies of this antibody fragment or in Part A of this study (i.e. the same patient cannot participate in Part A and B)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Local tolerability: Investigator's assessment of local tolerability using a validated score for each treatment area. Patient's assessment of subjective tolerability sensations (burning, itching, pain) recorded on a visual analogue scale (VAS) (0-10 | 28 days

SECONDARY OUTCOMES:
Safety variables: | 28 days
  Adverse events Detection of anti-drug antibodies (ADAs). Assessment of immunogenic potential of DLX105 by ELISA with coated DLX105 to capture anti-DLX105 antibodies
Efficacy variables | 28 days
  clinical signs of pharmacodynamic activity to intra-dermal administration of DLX105

CONTACTS AND LOCATIONS:
Locations (2):
- Universitätsklinikum, Vienna, Austria
- Universitätsklinikum Münster (UKM), Münster, Germany